CLINICAL TRIAL: NCT01569048
Title: Randomized Controlled Trial to Evaluate of Dexmedetomidine for the Effect on Operative Visibility in Patients Undergoing Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0023
Record Dates: First submitted 2012-03-23; First posted 2012-04-02 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Chronic Sinusitis
MeSH Terms: interventions — Propofol; Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- remifentanil (Active Comparator)
  Interventions: Drug: propofol and remifentanil
- dexmedetomidine (Experimental)
  Interventions: Drug: Propofol and dexmedetomidine

INTERVENTIONS:
Drug: Propofol and dexmedetomidine — Both group : propofol effect site TCI 2-4 mcg/ml, Remifentanil group : remifentanil effect site-TCI 2-4ng/ml Dexmedetomidine group: dexmedetomidine 0.5mcg/kg loading and 0.5mcg/kg/hr infusion
  Arms: dexmedetomidine
Drug: propofol and remifentanil — Both group : propofol effect site TCI 2-4 mcg/ml, Remifentanil group : remifentanil effect site-TCI 2-4ng/ml Dexmedetomidine group: dexmedetomidine 0.5mcg/kg loading and 0.5mcg/kg/hr infusion
  Arms: remifentanil

SUMMARY:
Various maneuvers are commonly used to achieve the ideal operative field necessary for successful endoscopic sinus surgery (ESS). Dexmedetomidine, a potent alpha2 adrenoceptor agonist which dose-dependently reduces arterial blood pressure and heart rate, decreases the hemodynamic and catecholamine response. And dexmedetomidine has an effect of peripheral vasoconstriction thus it is thus theologically appropriate for reducing bleeding during intranasal operation.

The aim of this study is to compare the effect of dexmedetomidine, an alpha2-adrenoreceptor agonist, on intraoperative bleeding, propofol requirement and postoperative profiles to remifentanil , an ultrashort-acting opioid.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅰ-Ⅱ
* Aged between 20 and 70 year
* General anesthesia for endoscopic sinus surgery

Exclusion Criteria:

* Body mass index >30
* Congestive heart failure, Sinus Bradycardia(<50 BPM), Uncontrolled hypertension,
* Coagulopathy
* Drug addiction
* Pregnancy
* Allergic fungal infection

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
surgical satisfaction about visibility of operative field | Within 1 day of endoscopic sinus surgery finish including dressing of surgical wound
  subjective satisfaction about visibility of operative field by surgeon/ numerous rating scale / 0: worst - 10:best

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea